CLINICAL TRIAL: NCT04370691
Title: JET Enhanced Thrombectomy Intervention Registry - JETi Registry
Brief Title: JETi Lower Extremity Arterial Thrombosis
Acronym: JETi
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10433
Record Dates: First submitted 2020-04-23; First posted 2020-05-01 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Arterial Thrombosis
Keywords: ABT-CIP-10433; Arterial Thrombosis; Lower Extremity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JETi™ Hydrodynamic Thrombectomy System: Subjects who were treated with JETi™ Hydrodynamic Thrombectomy System were included.
  Interventions: Device: JETi lower extremity arterial thrombosis

INTERVENTIONS:
Device: JETi lower extremity arterial thrombosis — The JETi System is is a hydro-mechanical aspiration system, intended for the removal of intravascular thrombus. The system comprises of the JETi Catheter (6F or 8F), JETi Pump Set, JETi Saline Drive Unit (SDU), JETi Accessory Cart, JETi Suction tubing and JETi Non-Sterile Canister Set. The JETi System is designed to continuously aspirate thrombotic material into the catheter, where a high-pressure stream of saline within the catheter tip macerates the thrombus as it is aspirated.

SUMMARY:
The JETi Registry is a prospective, single-arm, multi-center study to collect real-world data on the safety, performance, and clinical benefits of the JETi™ Hydrodynamic Thrombectomy System (JETi System) for the treatment of acute/subacute thrombosis in the peripheral vasculature. This post-market study will register approximately 280 subjects at approximately 30 centers Globally. Subjects participating in this Registry will be followed through their 12-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was treated or is expected to be treated for acute/subacute thrombosis, as determined by the investigator, in the peripheral vasculature with the JETi Hydrodynamic Thrombectomy System.
2. Subject or legally authorized representative must provide written informed consent.
3. Subject must be ≥ 18 years of age

Exclusion Criteria:

1. Subject has previously been registered in the JETi Registry in the last 12 months unless treated in the contralateral limb/different anatomy; patients treated in the contralateral limb/different anatomy within the last 12 months may re-enroll in the study.
2. Subject is currently participating in another drug or device clinical investigation.
3. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the past 20 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the patient population undergoing percutaneous treatment of thrombosis in the peripheral vascular system will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (21):
  - Honor Health, Scottsdale, Arizona
  - Arkansas Heart, Little Rock, Arkansas
  - PIH Good Samaritan, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University Hospital and Clinics, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - ClinRé, Thornton, Colorado
  - St. Mary Medical Center, Hobart, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Louisville, Louisville, Kentucky
  - Southoast Hospital, Fall River, Massachusetts
  - Henry Ford Detroit, Detroit, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Hendrick Medical Center, Abilene, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Charleston Area Medical Center, Charleston, West Virginia
- Royal Perth Hospital, Perth, Australia
- Hôpital Saint-François d'Assise, Québec, Quebec, Canada
- Germany (7):
  - University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Marien Hospital Herne, Herne, North Rhine-Westphalia
  - Klinikum Hochsauerland, Arnsberg
  - Evangelisches Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Sankt Gertrauden Krankenhaus, Berlin
  - Medizinische Einrichtungen der Universität zu Köln, Cologne
  - Universitätsklinikum Giessen, Giessen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 subjects with LEAT were registered across 18 sites: 62.0% (80/129) were from US sites, and 38.0% (49/129) were from non-US sites. At the time of data cut-off, all LEAT subjects had met the upper window of 30-day follow-up visit; 12-month follow-up visit is ongoing.
Groups:
- JETi™ Hydrodynamic Thrombectomy System: Subjects who were treated with JETi™ Hydrodynamic Thrombectomy System will be included.
  JETi lower extremity arterial thrombosis: The JETi System is is a hydro-mechanical aspiration system, intended for the removal of intravascular thrombus. The system comprises of the JETi Catheter (6F or 8F), JETi Pump Set, JETi Saline Drive Unit (SDU), JETi Accessory Cart, JETi Suction tubing and JETi Non-Sterile Canister Set. The JETi System is designed to continuously aspirate thrombotic material into the catheter, where a high-pressure stream of saline within the catheter tip macerates the thrombus as it is aspirated.
Period: Overall Study
Arm/Group | JETi™ Hydrodynamic Thrombectomy System
Started | 129
Completed | 42
Not Completed | 87
Not completed — Pending visit | 48
Not completed — Have Not Reached Lower Window | 15
Not completed — Termination | 14
Not completed — Missed or Overdue | 10

BASELINE CHARACTERISTICS:
Groups:
- JETi™ Hydrodynamic Thrombectomy System: JETi lower extremity arterial thrombosis: Subjects who were treated with JETi™Hydrodynamic Thrombectomy System will be included.
  The JETi System is is a hydro-mechanical aspiration system, intended for the removal of intravascular thrombus. The system comprises of the JETi Catheter (6F or 8F), JETi Pump Set, JETi Saline Drive Unit (SDU), JETi Accessory Cart, JETi Suction tubing and JETi Non-Sterile Canister Set. The JETi System is designed to continuously aspirate thrombotic material into the catheter, where a high-pressure stream of saline within the catheter tip macerates the thrombus as it is aspirated.
Arm/Group | JETi™ Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 64
  Others | 3
  Unknown or Not Reported | 50
Acute Limb Ischemia [Count of Participants; unit: Participants] | 68
Acute Limb Ischemia: In-Stent thrombosis [Count of Participants; unit: Participants] | 13
Acute Limb Ischemia: Acute graft thrombosis [Count of Participants; unit: Participants] | 12
Peripheral Artery Disease with Claudication (Rutherford 1-3) [Count of Participants; unit: Participants] | 15
Peripheral Artery Disease with CLTI (Rutherford 4-5) [Count of Participants; unit: Participants] | 21

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint - Clot Removal Grade From Pre-JETi to Post-JETi - Core Lab Assessed - Per Vessel Analysis
Description: Clot removal grade for each JETi-treated target vessel from pre-JETi angiogram to post-JETi angiogram (post-JETi thrombectomy and prior to any adjunctive therapies to treat underlying culprit lesions) per the grades. The independent imaging core laboratory will be responsible for assessing this endpoint.
  The rate of clot removal grade for each JETi-treated target vessel will be measured as per the Grades below:
  * Grade I: < 50% reduction
  * Grade II: 50- <95% reduction
  * Grade III: 95-100% reduction
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Units; unit: Vessels
Units Other Than Participants: Vessels
Groups:
- JETi™ Hydrodynamic Thrombectomy System: Subjects who were treated with JETi™Hydrodynamic Thrombectomy System will be included.
  The JETi System is is a hydro-mechanical aspiration system, intended for the removal of intravascular thrombus. The system comprises of the JETi Catheter (6F or 8F), JETi Pump Set, JETi Saline Drive Unit (SDU), JETi Accessory Cart, JETi Suction tubing and JETi Non-Sterile Canister Set. The JETi System is designed to continuously aspirate thrombotic material into the catheter, where a high-pressure stream of saline within the catheter tip macerates the thrombus as it is aspirated.
Arm/Group | JETi™ Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 122
Number analyzed (Vessels) | 129
Vessels
  Grade I | 36
  Grade II | 41
  Grade III | 52
  Grade II or Grade III | 93

2. Primary Outcome: Primary Safety Endpoint - Composite Rate of JETi-related MAEs
Description: JETi-related events defined as device-related death, major amputation of the treated limb, or major bleeding up to 30 days post-JETi procedure and as adjudicated by a clinical events committee (CEC).
Time Frame: Up to 30 days post-JETi procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | JETi™ Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 129
participants | 0 [0.00 to 2.82]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | JETi™ Hydrodynamic Thrombectomy System
All-Cause Mortality (participants affected / at risk) | 7/129
Serious Adverse Events (participants affected / at risk) | 28/129
Other Adverse Events (participants affected / at risk) | 16/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JETi™ Hydrodynamic Thrombectomy System (N=129)
Acute Myocardial Infarction (Cardiac disorders) | 1
Angina Unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 1
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1
Abdominal Hernia (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 3
Death (General disorders) | 5
Fatigue (General disorders) | 1
Abdominal Abscess (Infections and infestations) | 1
Coronavirus Infection (Infections and infestations) | 1
Diabetic Foot Infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Arterial Restenosis (Injury, poisoning and procedural complications) | 5
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Shunt Stenosis (Injury, poisoning and procedural complications) | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 3
Angiogram Peripheral (Investigations) | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Renal Artery Stenosis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1
Femoral Hernia Repair (Surgical and medical procedures) | 1
Foot Amputation (Surgical and medical procedures) | 2
Limb Amputation (Surgical and medical procedures) | 4
Peripheral Revascularisation (Surgical and medical procedures) | 2
Toe Amputation (Surgical and medical procedures) | 2
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 3
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
Peripheral Artery Occlusion (Vascular disorders) | 1
Peripheral Artery Stenosis (Vascular disorders) | 1
Peripheral Artery Thrombosis (Vascular disorders) | 8
Peripheral Embolism (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 5
Peripheral Vascular Disorder (Vascular disorders) | 2
Not Coded (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JETi™ Hydrodynamic Thrombectomy System (N=129)
Acute Myocardial Infarction (Cardiac disorders) | 0
Angina Unstable (Cardiac disorders) | 0
Arrhythmia (Cardiac disorders) | 0
Atrial Fibrillation (Cardiac disorders) | 0
Cardiac Failure (Cardiac disorders) | 0
Myocardial Infarction (Cardiac disorders) | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0
Abdominal Hernia (Gastrointestinal disorders) | 0
Abdominal Pain (Gastrointestinal disorders) | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0
Haematochezia (Gastrointestinal disorders) | 0
Chest Pain (General disorders) | 0
Death (General disorders) | 0
Fatigue (General disorders) | 0
Peripheral Swelling (General disorders) | 1
Abdominal Abscess (Infections and infestations) | 0
Cellulitis (Infections and infestations) | 1
Coronavirus Infection (Infections and infestations) | 0
Diabetic Foot Infection (Infections and infestations) | 0
Gangrene (Infections and infestations) | 0
Infection (Infections and infestations) | 0
Osteomyelitis (Infections and infestations) | 0
Pneumonia (Infections and infestations) | 0
Rectal Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 0
Vascular Access Site Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 0
Arterial Restenosis (Injury, poisoning and procedural complications) | 4
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0
Shunt Stenosis (Injury, poisoning and procedural complications) | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Angiogram Peripheral (Investigations) | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
Syncope (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0
Femoral Hernia Repair (Surgical and medical procedures) | 0
Foot Amputation (Surgical and medical procedures) | 0
Limb Amputation (Surgical and medical procedures) | 0
Peripheral Revascularisation (Surgical and medical procedures) | 0
Toe Amputation (Surgical and medical procedures) | 0
Haematoma (Vascular disorders) | 0
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0
Peripheral Artery Occlusion (Vascular disorders) | 0
Peripheral Artery Stenosis (Vascular disorders) | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1
Peripheral Embolism (Vascular disorders) | 0
Peripheral Ischaemia (Vascular disorders) | 0
Peripheral Vascular Disorder (Vascular disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Inst. may publish data/results individually from its site after any of (1) a multi-center publication is published, (2) no multicenter publication is submitted within 18months after closure of the Study, or (3) Abbott confirms there will be no multi-center publication. Inst. shall provide Sponsor with draft at least 60 days prior to submission for Sponsor review/comment. Upon request, Publication shall be delayed an additional 60 days. Due consideration will be given to Sponsor comments.

DOCUMENTS (2):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04370691/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04370691/SAP_001.pdf